CLINICAL TRIAL: NCT02567448
Title: Pathophysiology of the Upper Airway in Patients With Chronic Obstructive Pulmonary Disease (COPD) and Concomitant Obstructive Sleep Apnea (OSA)
Brief Title: Pathophysiology of the Upper Airway in Patients With COPD and Concomitant OSA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failed to accrue
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Robert L. Owens, Assistant Professor, University of California, San Diego
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UCSD130851
Record Dates: First submitted 2015-09-27; First posted 2015-10-05 (Estimated); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Chronic Obstructive Pulmonary Disease; Overlap syndrome; Pcrit; Critical closing pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive; Pulmonary Disease, Chronic Obstructive | interventions — Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- COPD Group (Active Comparator): Patients who were previously diagnosed of moderate to severe COPD as determined by spirometry. All patients will have sleep and pulmonary physiologic measurements.
  Interventions: Other: Sleep and pulmonary physiologic measurements
- Normal Control Group (Active Comparator): Patients who are healthy, without major medical or sleep problems, and have normal spirometry. All patients will have sleep and pulmonary physiologic measurements.
  Interventions: Other: Sleep and pulmonary physiologic measurements

INTERVENTIONS:
Other: Sleep and pulmonary physiologic measurements — Two overnight sleep studies, CT scan of upper airway and chest, pulmonary function test and pharyngeal lavage

SUMMARY:
The purpose of study is to evaluate the physiologic effects of pulmonary tissue/structural changes associated with COPD and upper airway inflammation on upper airway collapsibility. Upper airway collapsibility is closely associated with development of obstructive sleep apnea (OSA), which is a common disease characterized by repetitive collapse of upper airway during sleep, leading to hypoxemia and arousal. OSA has important neurocognitive and cardiovascular consequences, especially in patients with COPD.

Participants in this research study will undergo two overnight sleep studies (PSGs), pulmonary function test, and CT scan of the upper airway and chest. The first sleep study will evaluate the sleep breathing disorder and the second sleep study will measure the upper airway collapsibility, called critical closing pressure (Pcrit). Pcrit is measured by a modified continuous positive airway pressure (CPAP) machine which can provide a wide range of pressures between 20 and -20 cmH2O in order to modify upper airway pressure.

DETAILED DESCRIPTION:
This is a physiologic study to assess the effects of lower airway and lung tissue changes of COPD on upper airway collapsibility. Increased in lung volume and destruction of alveolar wall in COPD may have opposite and various effects on the upper airway collapsibility, which is an important factor of OSA development.

Chronic obstructive pulmonary disease (COPD) and obstructive sleep apnea (OSA) are very common disorders associated with considerable morbidity, mortality, and healthcare costs. The prevalence of both co-existing conditions is estimated to be ~4% of the general population. This COPD-OSA "overlap" syndrome causes more severe hypoxemia than either COPD or OSA alone and has important clinical consequences, including death. COPD is usually excluded in OSA research and OSA is typically excluded or not assessed in studies of COPD; thus, available information about the "overlap" syndrome is limited. Therefore, it is important to identify patients with both COPD and OSA and determine the mechanisms of poor outcomes for these patients in order to optimize therapy. The pathophysiology of the COPD-OSA syndrome is not well understood. The investigators propose to investigate upper airway (UA) anatomic characteristics and collapsibility as potential underlying mechanisms that may help to explain the negative additive effect of having both conditions. The objectives are to study CT measures of airway anatomy and the critical closing pressure of the upper airway (Pcrit), a gold standard measure of upper airway collapsibility, in patients with COPD-OSA compared with COPD only and normal controls. CT scan of upper airway and chest will allow precise measures of upper airway characteristics and COPD associated alveolar and lower airway ch. angesMeasures of upper airway collapsibility will provide us information about the mechanical nature of the airway and if the patients are more likely to have OSA. Subjects with COPD-OSA may exhibit more upper airway inflammation possibly due to their pre-existing COPD disease and the reoccurring opening and closing of the upper airway due to the OSA. Therefore the investigators would like to assess the degree of inflammation in these patients compared to normal controls.

ELIGIBILITY:
Inclusion Criteria for COPD Subjects:

* Age range 40-70 years.
* Demonstrated moderate to severe COPD as determined by spirometry (post-bronchodilator spirometry FEV1/FVC < 0.70 for diagnosing CODP and FEV1<80% predicted for staging)
* Smoking history of ≥ 10 pack-years

Inclusion Criteria for Control Subjects

* Age range 40-70 years
* Demonstrated no COPD as determined by normal spirometry (post-bronchodilator spirometry FEV1/FVC > 0.70 for diagnosing CODP and FEV1<80% predicted for staging)
* No smoking history as defined by less than 100 cigarettes smoked in a lifetime

Exclusion Criteria for both COPD and Control Subjects:

* Metal objects that may interfere with chest CT quantification including presence of a cardiac pacemaker, defibrillator, metal prosthetic heart valve, metal projectile or metal weapon fragment (bullet, shrapnel, shotgun shot) or metal shoulder prosthesis
* Subjects unable to perform spirometry due to:

  * chest or abdominal surgery in the past three months
  * a heart attack in the last three months
  * detached retina or eye surgery in the past three months
  * hospitalization for any other heart problem in the past month
* History of hypersensitivity to Afrin, Lidocaine or albuterol
* A psychiatric disorder, other than mild depression; e.g. schizophrenia, bipolar disorder, major depression, panic or anxiety disorders.
* More than 10 cups of beverages with caffeine (coffee, tea, soda/pop) per day
* Pregnancy or suspected pregnancy

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-08-11 (Actual); Study Completion 2016-08-11 (Actual)

PRIMARY OUTCOMES:
Critical closing pressure (PCrit) | Baseline
  Measured during overnight sleep study

SECONDARY OUTCOMES:
Pharyngeal lavage cell count distribution | Baseline
Minimal later airway dimension (mLAT) | Baseline
  Measured from upper airway CT scan
Minimal anteroposterior airway dimension (mAP) | Baseline
  Measured from upper airway CT scan
Minimal cross sectional airway area (mCSA) | Baseline
  Measured from upper airway CT scan
Lateral airway dimension on hard palate/uvula/epiglottis level | Baseline
  Measured from upper airway CT scan
Anteroposterior airway dimension on hard palate/uvula/epiglottis level | Baseline
  Measured from upper airway CT scan
Cross-sectional airway area on hard palate/uvula/epiglottis level | Baseline
  Measured from upper airway CT scan
Distance between the lower edge of the mandible and the lower edge of the hyoid (MH) | Baseline
  Measured from upper airway CT scan
Upper airway length | Baseline
  Measured from upper airway CT scan
Width of hard palate | Baseline
  Measured from upper airway CT scan
Nasophayngeal/retropalatal/retroglossal pharyngeal cavity volume | Baseline
  Measured from upper airway CT scan
Volume within the cervico-mandibular bony frame | Baseline
  Measured from upper airway CT scan
Volume of retropalatal/retroglossal soft tissue | Baseline
Parapharyngeal fat pad volume | Baseline
Tongue volume | Baseline
Emphysema score | Baseline
  Measured from CT chest scan
Emphysema distribution | Baseline
  Measured from CT chest scan
Lower airway wall thickness on chest CT scan | Baseline
  Measured from CT chest scan
Forced expiratory volume in 1 second (FEV1) | Baseline
Total lung capacity (TLC) | Baseline
Ratio of residual volume / total lung capacity (RV/TLC) | Baseline
Diffusing capacity of the lung for carbon monoxide (DLCO) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Soler, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States